CLINICAL TRIAL: NCT05033366
Title: Relationship Between Fertility Hormone Patterns and Pregnancy Rates.
Status: Enrolling by invitation | Type: Observational
Sponsor: MFB Fertility (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021/03/29
Record Dates: First submitted 2021-07-30; First posted 2021-09-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related; Hormone Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Proov test strip users that record results with the Proov app: Participants using Proov test strips along with the Proov app who have logged at least one complete cycle will be asked to complete an online survey about fertility test results and current/previous pregnancy status. They will also be asked cycle history (irregular vs regular, cycle length), fertility testing (partners semen analysis results, AMH level, HSG results), possible fertility medications taken or prescribed, age, race, smoking status, and BMI.
  Interventions: Diagnostic Test: Proov Test

INTERVENTIONS:
Diagnostic Test: Proov Test — Rapid response urine PdG, FSH, E1G and LH test strips, Proov

SUMMARY:
The purpose of this study is to determine if certain patterns of hormone levels during the menstrual cycle are correlated with different pregnancy outcomes.

DETAILED DESCRIPTION:
Proov tests are fertility tracking tests. They are used for monitoring ovulation at home, and are able to measure one or more hormones. These hormones can predict and confirm ovulation. Tracking these hormones can help a woman understand if she is ovulating, and can help to identify problems that could be preventing pregnancy.

After giving permission to access your testing history collected in the Proov app from March 2020 to April 2022, you will complete an online survey about your fertility test results and pregnancy status. You will also be asked information regarding your age, race, smoking status, and BMI. Your test results logged in the Proov app will be shared automatically. You will need 10-20 minutes to fill out the fertility survey.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 18 - no limit
3. Have completed one full cycle using the Proov app

Exclusion Criteria:

1. Male
2. Have not completed one full cycle using the Proov app

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Females age 18 - no limit who are using, or have used, the Proov hormone test strips and the Proov app for at least one full cycle.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
self reported pregnancy | Two menstrual cycle, up to 45 days each
  Questionnaire used to assess if positive Proov test strips measuring urine PDG correlate with increased rates of self reported pregnancy

SECONDARY OUTCOMES:
self reported first trimester pregnancy loss | Three months
  Questionnaire used to assess if negative Proov test strips measuring urine PDG correlate with increased rates of self reported first trimester pregnancy loss

CONTACTS AND LOCATIONS:
Overall Officials: Amy Beckely, PhD, Principal Investigator — MFB Fertility
Locations (1):
- MFB Fertility, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
only cohort data will be released